CLINICAL TRIAL: NCT01504750
Title: Healing Patient Rooms; The Effect of Lighting on Recovery and Well-being of Patients
Brief Title: Healing Patient Rooms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Philips Lighting Eindhoven (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GOAL/HH/014/2009
Record Dates: First submitted 2011-11-14; First posted 2012-01-05 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Depression; Headache; Sleep
Keywords: Length of Stay [E02.760.400.480]; Activities of Daily Living [I03.050]
MeSH Terms: conditions — Depression; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lighting room (Experimental): In the ceiling, luminaires are installed that offer the basic lighting in the patient room that will automatically and gradually change in light level (100-300 lux) and color temperature (3000-4000 K). This so called daily rhythm light meets the EN12464-1 standard for patient rooms in hospitals.
  Interventions: Procedure: dynamic daylight and atmosphere lighting
- control room (No Intervention): Normal lighted patient room

INTERVENTIONS:
Procedure: dynamic daylight and atmosphere lighting — In the ceiling, luminaires are installed that offer the basic lighting in the patient room that will automatically and gradually change in light level (100-300 lux) and color temperature (3000-4000 K). This so called daily rhythm light meets the EN12464-1 standard for patient rooms in hospitals. The system offers a light boost by bringing the illuminance to a level of maximal 2000 lux and 7000 K, during a period of two hours in the morning. Besides, a low intensity color cove as well as some white LED spots are added to create a pleasant ambience in the patient room. The illuminance is between 50 and 60 lux and, depending on the color choice, the color temperature is 2300 K (relax) or 3800 K (active). The lighting solution used is HealWell of Philips Lighting.
  Arms: lighting room

SUMMARY:
Rationale:

Many study reports described benefits of natural sunlight. It is believed that artificial light can achieve similar benefits as sunlight and can be used to compensate for the lack of sunlight, for instance in north-facing hospital rooms or during wintertime.

The most plausible paths mediating the effects of light are:

* the biological effect of light, relating to circadian biology and the sleep/wake-rhythm;
* the emotional/psychological effects of light, relating to mood/stress and the antidepressant action of light .

Objective:

The project aims to measure, evaluate and quantify the beneficial effects of a dynamic daylight & atmosphere experience in patient rooms for cardiovascular patients during the dark months of the year.

Study design:

The study involves an experiment in which psychological, emotional and clinical parameters of patients in hospital rooms with standard light situation are compared with those of patients in rooms with a dynamic daylight & atmosphere experience.

Study population:

The population includes cardiovascular patients who reside in the general cardiology department of the Maastricht University Hospital (18 patient beds) with an intended minimum length of stay of 3 days, who have given written consent.

Intervention:

Half of the patient rooms on the ward are equipped with special luminaires. In the ceiling, luminaires are installed that offer the basic lighting in the patient room that will automatically and gradually change in light level (100-300 lux) and color temperature (3000-4000 K). This so called daily rhythm light meets the EN12464-1 standard for patient rooms in hospitals. The same luminaires in the ceiling will also offer the light boost by bringing the illuminance to a level of maximal 2000 lux and 7000 K, during a period of two hours in the morning. Besides the ceiling luminaires, a low intensity color cove as well as some white LED spots are added to create a pleasant ambience in the patient room

Main study parameters/endpoints:

The primary study measures are length of stay and quality of recovery expressed by physiological, emotional and clinical parameters. Also the effect on patient satisfaction is determined using pre and post assessments.

DETAILED DESCRIPTION:
Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Regular measurements for patient care will be mainly used as outcome measures. Some of the psychological parameters are measured in regular care (e.g. pain score). Other psychological parameters will be measured with an additional questionnaire (depression, appetite, delirium, sleep quality and sleepiness). A trained research nurse will visit all participating patients in their rooms to assist with completing the questionnaires. This way of data collection will pose a minimal burden on the patients (maximum 30 minutes on daily basis). The risks of the intervention are negligible, because the light level will not exceed outside luminance on a cloudy day and meets all CIE safety standards (ref. CIE S009).

ELIGIBILITY:
Inclusion Criteria:

- patients admitted to study room

Exclusion Criteria:

* Age under 18 years
* Blindness
* Unability to obtain informed consent
* Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Length of stay | participants will be followed for the duration of their stay at the cardiology ward (an expected average of 6 days) and one week thereafter
  Does a dynamic daylight & atmosphere experience improve the recovery of cardiovascular patients expressed in length of stay.

SECONDARY OUTCOMES:
general well-being | participants will be followed for the duration of their stay at the cardiology ward (an expected average of 6 days) and two weeks thereafter
  Does a dynamic daylight & atmosphere experience increase the general well-being (sleepiness/alertness, cognitive functioning, sleep quality and appetite) and satisfaction of cardiovascular patients?

CONTACTS AND LOCATIONS:
Overall Officials: Petra Kuijpers, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands